CLINICAL TRIAL: NCT06549361
Title: The Retrospective Clinical Study of Extranodal Diffuse Large B-Cell Lymphoma
Brief Title: A Retrospective Study on Extranodal DLBCL
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Other Study IDs: ENI-DLBCL
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma; Extranodal Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: Lymphoma; Extranodal
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions need to be specified for this study — No interventions need to be specified for this study

SUMMARY:
The aim of this study is to prospectively collect clinical information of patients with extranodal DLBCL, assess the effectiveness of treatment for extranodal DLBCL in the real world, and explore the optimal treatment strategies in real-world populations.

DETAILED DESCRIPTION:
DLBCL is a highly common aggressive non-Hodgkin's lymphoma. For specific extranodal sites of DLBCL, traditional chemotherapy protocols often cannot provide satisfactory results for patients. The aim of this study is to prospectively collect clinical information of patients with extranodal DLBCL, including the distribution of involved sites (such as central nervous system, testes, skin, breast, gastrointestinal tract, etc.), prognosis of diffuse large B-cell lymphoma with involvement of different extranodal sites, genetic mutation characteristics, correlation with molecular subtypes, impact of different treatment regimens on efficacy, assess the effectiveness of treatment for extranodal DLBCL in the real world, and explore the optimal treatment strategies in real-world populations.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥ 18 years (including 18 years).
* 2. Pathologically diagnosed with diffuse large B-cell lymphoma according to the 2016 WHO classification, including non-specific types and various special subtypes.
* 3. Newly diagnosed DLBCL with involvement of extranodal organs.
* 4. Patients who have received clinical treatment for lymphoma.
* 5.Patients with measurable lesions, including at least one effective efficacy assessment.

Exclusion Criteria:

* 1. Patients receiving supportive care only.
* 2. Patients who cannot obtain effective efficacy assessment data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically confirmed diagnosis of non-Hodgkin lymphoma with extranodal involvement or non-Hodgkin lymphoma of rare pathological types attending participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 5023 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Time Frame: Baseline up to data cut-off (up to approximately 1 year)
  Overall Survival (OS) will be defined from the start date of therapy to the date of death from any cause.
Progression Free Survival (PFS) | Time Frame: Baseline up to data cut-off (up to approximately 1 year)
  Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.

SECONDARY OUTCOMES:
Clinical characteristics form | Baseline up to data cut-off (up to approximately 1 year)
  Clinical characteristics from data filled into registry forms by physicians and data managers, including but not limited to values of lactate dehydrogenase, clinical stage, performance status, age ≥ 60 years and number and location of extranodal localizations.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China